CLINICAL TRIAL: NCT03575260
Title: 500mg Fulvestrant Versus Exemestane in Metastatic Breast Cancer (MBC) Resistant to Adjuvant Non-steroidal Aromatase Inhibitors in Clinical Practice- a Multicenter Retrospective Study
Brief Title: 500mg Fulvestrant Versus Exemestane in MBC
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-2
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: Fulvestrant; Exemestane
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fulvestrant: Fulvestrant 500 mg on days 0, 14, and 28, and every 28 days thereafter
- Exemestane: Exemestane 25mg per day

SUMMARY:
500mg Fulvestrant versus Exemestane in MBC

DETAILED DESCRIPTION:
500mg Fulvestrant versus Exemestane in Metastatic Breast Cancer (MBC) resistant to adjuvant Non-steroidal Aromatase Inhibitors in clinical practice- a multicenter retrospective study

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman, age > 18 years old
* Diagnosed with ER/PR+，HER2- Metastatic Breast Cancer
* Adjuvant treatment of Non-steroidal Aromatase Inhibitors
* First line of Metastatic Breast Cancer is 500mg Fulvestrant or Exemestane for at least one month, starting from 2014.01.01-2017.06.01
* Available medical history

Exclusion Criteria:

* Incomplete medical history

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Biyun Wang, MD, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xie Y, Li Y, Zhang Y, Zhang S, Li W, Guan X, Zhao Y, Gong C, Hu X, Zhang J, Cao E, Wang L, Ge R, Wang B. Fulvestrant 500 mg Versus Exemestane in Postmenopausal Women With Metastatic Breast Cancer Resistant to Adjuvant Nonsteroidal Aromatase Inhibitors in Clinical Practice: A Multicenter Retrospective Study. Clin Breast Cancer. 2019 Jun;19(3):e452-e458. doi: 10.1016/j.clbc.2019.01.015. Epub 2019 Feb 7. PMID 30846408